CLINICAL TRIAL: NCT06451471
Title: Assessment of Serum Galectin-3 Level as an Indicator of Subclinical Inflammation in Patients With Familial Mediterranean Fever
Brief Title: "Galectin-3 as a Marker of Subclinical Inflammation in FMF"
Status: Completed | Type: Observational
Sponsor: Turkish League Against Rheumatism (Other)
Responsible Party: Principal Investigator, Oguzhan Lacin, Medical Doctor, Turkish League Against Rheumatism
Other Study IDs: TRASD-OL-TEZ
Record Dates: First submitted 2024-06-04; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Ailesel Akdeniz Ateşi
Keywords: GALEKTİN-3; Subclinical Inflammation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Active Comparator: Group 1: PATIENT GROUP DIAGNOSED WITH FMF
- Active Comparator: Group 2: HEALTHY CONTROL GROUP

SUMMARY:
The goal of this observational study is to learn about the relationship between serum Galectin-3 levels and subclinical inflammation in patients with Familial Mediterranean Fever (FMF). The main questions it aims to answer are:

* Are serum Galectin-3 levels higher in FMF patients compared to healthy controls?
* Is there a positive correlation between serum Galectin-3 levels and Serum Amyloid A (SAA) protein levels in FMF patients?

Participants will:

* Provide blood samples to measure serum Galectin-3 and SAA levels.
* Complete a sociodemographic and clinical data form.
* Fill out the FMF Quality of Life (QoL) scale.

Researchers will compare FMF patients and healthy controls to see if there are significant differences in serum Galectin-3 levels and to determine the correlation between Galectin-3 and SAA protein levels in FMF patients.

ELIGIBILITY:
Inclusion Criteria:

* for the Patient Group:

  1. Aged between 18 and 65 years,
  2. Able to provide written informed consent for the study,
  3. Literate,
  4. Diagnosed with Familial Mediterranean Fever (FMF) according to the Tel Hashomer criteria and not currently experiencing an attack (with at least 15 days since the last attack).

     * Inclusion Criteria for the Healthy Control Group:

  <!-- -->

  1. Aged between 18 and 65 years,
  2. Able to provide written informed consent for the study,
  3. Literate.

Exclusion Criteria:

* Exclusion Criteria for the Patient Group:

  1. Presence of known inflammatory diseases other than FMF,
  2. Presence of known systemic, chronic, severe medical conditions,
  3. Presence of active infection,
  4. Conditions affecting cognitive functions such as mental retardation, delirium, dementia, epilepsy, and alcohol or substance use disorders,
  5. Being pregnant or in the lactation period.
* Exclusion Criteria for the Healthy Control Group:

  1. Presence of known systemic, chronic, severe medical conditions,
  2. Presence of inflammatory diseases,
  3. Presence of active infection,
  4. Conditions affecting cognitive functions such as mental retardation, delirium, dementia, epilepsy, and alcohol or substance use disorders,
  5. Being pregnant or in the lactation period. -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Aged between 18 and 65 years,
  2. Able to provide written informed consent for the study,
  3. Literate,
  4. Diagnosed with Familial Mediterranean Fever (FMF) according to the Tel Hashomer criteria and not currently experiencing an attack (with at least 15 days since the last attack).
Sampling Method: Non-Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Serum Galectin-3 Levels | 2022
  Comparison of serum Galectin-3 levels between FMF patients and healthy controls to determine if there is a significant difference.

SECONDARY OUTCOMES:
Serum Amyloid A (SAA) Levels | 2022
  Measurement of SAA levels in both FMF patients and healthy controls.
Correlation Analysis | 2022
  Determination of the correlation between serum Galectin-3 levels and SAA levels in FMF patients.
Clinical Variables | 2022
  Analysis of the relationship between Galectin-3/SAA levels and clinical variables such as age, BMI, disease duration, and frequency of FMF attacks.

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University Faculty of Medicine, Erzurum, Turkey (Türkiye)